CLINICAL TRIAL: NCT01675154
Title: Phase 2 Study of Orlistat and SLx-4090 for the Treatment of Type 1 Hyperlipoproteinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to unavailability of the drug.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abhimanyu Garg, PI, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3940; FD-R-003940
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Type 1 Hyperlipoproteinemia
Keywords: hypertriglyceridemia
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome; Hypertriglyceridemia | interventions — Orlistat; 6-(4'-trifluoromethyl-6-methoxybiphenyl-2-ylcarboxamido)-1,2,3,4-tetrahydroisoquinoline-2-carboxylic acid phenyl ester

STUDY DESIGN:
Intervention Model Description: This trial is adaptive design/flexible design. The participants were randomized from the start of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SLx-4090 placebo/Orlistat Placebo (Placebo Comparator): Slx-4090(placebo) is dosed as 4 tablets of 50 mg, three times per day with meals.
  Orlistat (placebo) is dosed as 2 capsules of 60 mg, three times per day with meals.
  This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
  Interventions: Drug: SLx-4090 placebo; Drug: Orlistat Placebo
- Orlistat/placebo (Experimental): Orlistat two capsules 60mg each, three times per day with meals. Placebo for SLx-4090, 4 tablets 50mg each, three times per day with meals. This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
  Interventions: Drug: SLx-4090 placebo; Drug: Orlistat
- Orlistat placebo /SLx-4090 (Experimental): Orlistat placebo 2 capsules, 60mg each three times per day with meals. Slx-4090 4 tablets, 50mg each. three times per day with meals. This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
  Interventions: Drug: Orlistat Placebo; Drug: Slx-4090
- Orlistat/SLx-4090 (Experimental): Orlistat, 2 capsules 60 mg each, three times per day with meals. SLx-4090 4 tablets 50mg each, three times per day with meals. This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
  Interventions: Drug: Orlistat; Drug: Slx-4090

INTERVENTIONS:
Drug: SLx-4090 placebo — Given for 4 weeks
  Arms: Orlistat/placebo; SLx-4090 placebo/Orlistat Placebo
Drug: Orlistat Placebo — Given for 4 weeks
  Arms: Orlistat placebo /SLx-4090; SLx-4090 placebo/Orlistat Placebo
Drug: Orlistat — Given for 4 weeks
  Arms: Orlistat/SLx-4090; Orlistat/placebo
Drug: Slx-4090 — Given for 4 weeks
  Arms: Orlistat placebo /SLx-4090; Orlistat/SLx-4090

SUMMARY:
Funding Source - FDA OOPD

This study is being done to find out whether an investigational (not approved by FDA ) drug called SLx-4090 or Orlistat (FDA approved medication for weight loss) when given alone or in combination can treat the high blood fat (elevated triglycerides)levels found in the condition Type 1 Hyperlipoproteinemia (T1HLP) better or more safely than low fat diet alone, the current standard medical care.

It is also not clear whether Orlistat, that is FDA approved for weight loss, is effective in lowering blood fat levels in patients with Type 1 hyperlipoproteinemia (T1HLP). The researchers are interested in learning whether any one of these drugs when given alone or in combination is more effective and safe in treating T1HLP.

DETAILED DESCRIPTION:
Type I hyperlipoproteinemia is a rare, autosomal recessive metabolic disorder characterized by extreme hypertriglyceridemia due to a deficiency in lipoprotein lipase or related proteins. Treatment of these patients is challenging as triglyceride-lowering medications are ineffective. A low fat diet is helpful, however, despite good dietary compliance, some patients continue to have severe hypertriglyceridemia and recurrent pancreatitis which can be life threatening. Therefore, we wish to investigate whether inducing dietary fat malabsorption or inhibiting chylomicron formation will cause further lowering of serum triglycerides (TG) beyond the effect of limiting dietary fat intake.

We will study the efficacy and safety of an inhibitor of intestinal lipase (Orlistat) and an intestinal-specific inhibitor of microsomal triglyceride transport protein (MTP) involved in the assembly and secretion of chylomicrons (SLx-4090), alone and in combination, for reducing serum triglyceride levels in patients with Type I hyperlipoproteinemia. We plan to enroll 20 patients with Type I hyperlipoproteinemia in a randomized, double-blind, placebo-controlled, cross-over trial. After a baseline evaluation, the subjects will be randomly assigned to placebo/placebo, Orlistat/placebo, SLx-4090/placebo or Orlistat/SLx-4090 for the duration of four weeks followed by a one week wash out period. During the last week of each study period, fasting blood samples will be drawn for three consecutive days for serum lipids and chemistry panel. The primary endpoint will be serum triglycerides; the secondary endpoint variables will be fasting and postprandial serum chylomicron-TG levels, postprandial serum TG levels during a meal tolerance test and retinyl palmitate levels during a meal tolerance test. Repeated measures analysis of variance will be used for statistical comparisons.

Our results may help in designing novel therapeutic approaches for patients with Type 1 hyperlipoproteinemia.

ELIGIBILITY:
Inclusion Criteria:

* Type I hyperlipoproteinemia.
* Fasting serum triglyceride levels of greater than 1000 mg/dL.
* Age > 12 years

Exclusion Criteria:

* Secondary hypertriglyceridemias due to diabetes, renal disease, hypothyroidism, alcoholism and drug therapy such as estrogens and estrogen analogues, steroids, HIV-protease inhibitors, retinoic acid derivatives and interferons.
* Pregnant or lactating women
* Significant liver disease (elevated transaminases > 2 times upper limit of normal)
* Alcohol abuse (> 7 drinks or 84 g per week for women and > 14 drinks for men or 168 g per week for men)
* Drug use (cocaine, marijuana, LSD, etc.)
* Major surgery in the past three months
* Congestive heart failure
* Serum creatinine greater than 2.5 mg/dL
* Cancer within the past five years
* Gastrointestinal surgery in the past
* Current therapy with anti-coagulants, digoxin and anti-arrhythmics
* Chronic malabsorption syndromes
* Cholestasis
* Acute illnesses such as acute pancreatitis in the last 8 weeks

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - UT Southwestern Medical Center 5323 Harry Hines Blvd, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial is adaptive design/flexible design. The participants were randomized from the start of the study
Groups:
- SLx-4090 Placebo/Orlistat Placebo First: First, SLx-4090 (placebo) is dosed as 4 tablets of 50 mg, three times per day with meals.
  Orlistat (placebo) is dosed as 2 capsules of 60 mg, three times per day with meals.
  SLx-4090 placebo: Given for 4 weeks
  Orlistat Placebo: Given for 4 weeks
- Orlistat/SLx-4090 Placebo: Then, Orlistat two capsules 60 mg each, three times per day with meals. Placebo for SLx-4090, 4 tablets 50 mg each, three times per day with meals were administered
  SLx-4090 placebo: Given for 4 weeks
  Orlistat: Given for 4 weeks
- Orlistat Placebo /SLx-4090: Then, Orlistat placebo 2 capsules, 60 mg each three times per day with meals. SLx-4090 4 tablets, 50 mg each. three times per day with meals were administered
  Orlistat Placebo: Given for 4 weeks
  SLx-4090: Given for 4 weeks
- Orlistat/SLx-4090: Then, Orlistat, 2 capsules 60 mg each, three times per day with meals. SLx-4090 4 tablets 50 mg each, three times per day with meals were administered
  Orlistat: Given for 4 weeks
  SLx-4090: Given for 4 weeks
Period: First Intervention Period (4 Weeks)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: First Washout Period (1 Week)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started | 2 (Subjects were enrolled Regimen 1) | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention Period (4 Weeks)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started | 1 | 1 (Subjects were enrolled in Regimen 2) | 1 | 2
Completed | 0 | 1 | 1 | 1
Not Completed | 1 | 0 | 0 | 1
Period: Second Washout Period (1 Week)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started | 1 | 1 | 1 | 2
Completed | 1 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention Period (4 Weeks)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started (Further participation of two patients was halted after Period 2 due to unavailability of the study medications.) | 1 | 1 | 1 | 0
Completed | 1 | 0 | 1 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Third Washout Period (1 Week)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started | 1 | 0 | 1 | 0
Completed | 1 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention Period (4 Weeks)
Arm/Group | SLx-4090 Placebo/Orlistat Placebo First | Orlistat/SLx-4090 Placebo | Orlistat Placebo /SLx-4090 | Orlistat/SLx-4090
Started | 1 | 0 | 1 | 0
Completed (One patient dropped out during Period 3 due to personal reasons. Therefore, not included in this intervention period.) | 1 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are based on first intervention period assignment. This trial is an adaptive design/flexible design using responsive adaptive randomization. The participants were randomized from the start of the study
Groups:
- Placebo/Placebo at First Intervention Period: Slx-4090(placebo) is dosed as 4 tablets of 50 mg, three times per day with meals.
  Orlistat (placebo) is dosed as 2 capsules of 60 mg, three times per day with meals.
- Orlistat/Placebo at First Intervention Period: Orlistat two capsules 60mg each, three times per day with meals. Placebo for SLx-4090, 4 tablets 50mg each, three times per day with meals were administered.
- Orlistat Placebo /Slx-4090 at First Intervention Period: Orlistat placebo 2 capsules, 60mg each three times per day with meals. Slx-4090 4 tablets, 50mg each. three times per day with meals were administered
- Orlistat/SLx-4090 at First Intervention Period: Orlistat, 2 capsules 60 mg each, three times per day with meals. SLx-4090 4 tablets 50mg each, three times per day with meals were administered.
- Total: Total of all reporting groups
Arm/Group | Placebo/Placebo at First Intervention Period | Orlistat/Placebo at First Intervention Period | Orlistat Placebo /Slx-4090 at First Intervention Period | Orlistat/SLx-4090 at First Intervention Period | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 1 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2
  Male | 2 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 0 | 3
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Number; unit: participants]
  <18.5 kg/m^2 | 0 | 0 | 0 | 0 | 0
  18.5 kg/m^2-24.9 kg/m^2 | 1 | 0 | 0 | 1 | 2
  25 kg/m^2-29.9 kg/m^2 | 1 | 0 | 0 | 0 | 1
  30 kg/m^2-34.9 kg/m^2 | 0 | 1 | 1 | 0 | 2
  35 kg/m^2-39.9 kg/m^2 | 0 | 0 | 0 | 0 | 0
  >=40 kg/m^2 | 0 | 0 | 0 | 0 | 0
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 1969 (419) | 4840 (0) | 814 (0) | 2061 (0) | 2421 (1480)

OUTCOME MEASURES:

1. Primary Outcome: Serum Triglycerides at First Intervention Period
Description: Serum triglyceride level will be measured after taking each assigned intervention at first intervention period.
Time Frame: 4 weeks after the assigned treatment (first intervention period)
Population: This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- SLx-4090 Placebo/Orlistat Placebo: Slx-4090(placebo) is dosed as 4 tablets of 50 mg, three times per day with meals.
  Orlistat (placebo) is dosed as 2 capsules of 60 mg, three times per day with meals.
  SLx-4090 placebo: Given for 4 weeks
  Orlistat Placebo: Given for 4 weeks
- Orlistat/Placebo: Orlistat two capsules 60mg each, three times per day with meals. Placebo for SLx-4090, 4 tablets 50mg each, three times per day with meals.
  SLx-4090 placebo: Given for 4 weeks
  Orlistat: Given for 4 weeks
- Orlistat Placebo /Slx-4090: Orlistat placebo 2 capsules, 60mg each three times per day with meals. Slx-4090 4 tablets, 50mg each. three times per day with meals.
  Orlistat Placebo: Given for 4 weeks
  Slx-4090: Given for 4 weeks
- Orlistat/SLx-4090: Orlistat, 2 capsules 60 mg each, three times per day with meals. SLx-4090 4 tablets 50mg each, three times per day with meals.
  Orlistat: Given for 4 weeks
  Slx-4090: Given for 4 weeks
Arm/Group | SLx-4090 Placebo/Orlistat Placebo | Orlistat/Placebo | Orlistat Placebo /Slx-4090 | Orlistat/SLx-4090
Number analyzed (Participants) | 2 | 1 | 1 | 1
mg/dL | 2086 (481.54) | 3320 | 1576 | 1280

2. Primary Outcome: Serum Triglycerides at Second Intervention Period
Description: Serum triglyceride level will be measured after taking each assigned intervention at second intervention period
Time Frame: 4 weeks after the assigned treatment (Second Intervention Period)
Population: Patient assigned to SLX-4090 placebo/Orlistat placebo group withdrew from the study in this phase.
  One more subject was assigned to the Orlistat/SLx-4090 but could not start the study as the drug SLx-4090 was not available.
  This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SLx-4090 Placebo/Orlistat Placebo | Orlistat/Placebo | Orlistat Placebo /Slx-4090 | Orlistat/SLx-4090
Number analyzed (Participants) | 0 | 1 | 1 | 1
mg/dL |  | 1419 | 2040 | 3478

3. Primary Outcome: Serum Triglycerides at Third Intervention Period
Description: Serum triglyceride level will be measured after taking each assigned intervention at intervention period
Time Frame: 4 weeks after the assigned treatment (Third Intervention Period)
Population: Patient assigned to Orlistat/SLX-4090 placebo group did not start the assigned treatment due to lack of drugs.
  This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SLx-4090 Placebo/Orlistat Placebo | Orlistat/Placebo | Orlistat Placebo /Slx-4090 | Orlistat/SLx-4090
Number analyzed (Participants) | 1 | 0 | 1 | 0
mg/dL | 6220 |  | 1320 |

4. Primary Outcome: Serum Triglycerides at Fourth Intervention Period
Description: Serum triglyceride level will be measured after taking each assigned intervention at fourth intervention period
Time Frame: 4 weeks after the assigned treatment (Fourth Intervention Period)
Population: Patient assigned to Orlistat/SLX-4090 group did not start the assigned treatment due to lack of drugs.
  This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SLx-4090 Placebo/Orlistat Placebo | Orlistat/Placebo | Orlistat Placebo /Slx-4090 | Orlistat/SLx-4090
Number analyzed (Participants) | 1 | 0 | 1 | 0
mg/dL | 1156 |  | 2946 |

ADVERSE EVENTS:
Time Frame: Over a period of 1 year .
Description: This trial is adaptive design/flexible design. The participants were either randomized from the start of the study or after the completion of each treatment.
  Includes all participants who started first, second, third and fourth intervention periods. Events were collected separately for each period.
Groups:
- 1st Intervention Period:SLx-4090 Placebo/Orlistat Placebo; 2nd Intervention Period:SLx-4090 Placebo/Orlistat Placebo; 3rd Intervention Period:SLx-4090 Placebo/Orlistat Placebo; 4th Intervention Period:SLx-4090 Placebo/Orlistat Placebo: Slx-4090(placebo) is dosed as 4 tablets of 50 mg, three times per day with meals.
  Orlistat (placebo) is dosed as 2 capsules of 60 mg, three times per day with meals.
  SLx-4090 placebo: Given for 4 weeks
  Orlistat Placebo: Given for 4 weeks
- 1st Intervention Period:Orlistat/Placebo; 2nd Intervention Period:Orlistat/Placebo; 3rd Intervention Period:Orlistat/Placebo; 4th Intervention Period:Orlistat/Placebo: Orlistat two capsules 60mg each, three times per day with meals. Placebo for SLx-4090, 4 tablets 50mg each, three times per day with meals.
  SLx-4090 placebo: Given for 4 weeks
  Orlistat: Given for 4 weeks
- 1st Intervention Period:Orlistat Placebo /Slx-4090: Orlistat placebo 2 capsules, 60mg each three times per day with meals. Slx-4090 4 tablets, 50mg each. three times per day with meals.
  Orlistat Placebo: Given for 4 weeks
  Slx-4090: Given for 4 weeks
- 1st Intervention Period:Orlistat/SLx-4090; 2nd Intervention Period:Orlistat Placebo /Slx-4090; 2nd Intervention Period:Orlistat/SLx-4090; 3rd Intervention Period:Orlistat Placebo /Slx-4090; 3rd Intervention Period:Orlistat/SLx-4090; 4th Intervention Period:Orlistat Placebo /Slx-4090; 4th Intervention Period:Orlistat/SLx-4090: Orlistat, 2 capsules 60 mg each, three times per day with meals. SLx-4090 4 tablets 50mg each, three times per day with meals.
  Orlistat: Given for 4 weeks
  Slx-4090: Given for 4 weeks
Arm/Group | 1st Intervention Period:SLx-4090 Placebo/Orlistat Placebo | 1st Intervention Period:Orlistat/Placebo | 1st Intervention Period:Orlistat Placebo /Slx-4090 | 1st Intervention Period:Orlistat/SLx-4090 | 2nd Intervention Period:SLx-4090 Placebo/Orlistat Placebo | 2nd Intervention Period:Orlistat/Placebo | 2nd Intervention Period:Orlistat Placebo /Slx-4090 | 2nd Intervention Period:Orlistat/SLx-4090 | 3rd Intervention Period:SLx-4090 Placebo/Orlistat Placebo | 3rd Intervention Period:Orlistat/Placebo | 3rd Intervention Period:Orlistat Placebo /Slx-4090 | 3rd Intervention Period:Orlistat/SLx-4090 | 4th Intervention Period:SLx-4090 Placebo/Orlistat Placebo | 4th Intervention Period:Orlistat/Placebo | 4th Intervention Period:Orlistat Placebo /Slx-4090 | 4th Intervention Period:Orlistat/SLx-4090
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/0 | 0/1 | 0/0 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 1/2 | 0/1 | 0/1 | 0/1 | 0/0 | 0/1 | 0/0 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 1/1 | 1/1 | 1/1 | 0/1 | 0/1 | 1/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/0 | 0/1 | 0/0 | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=2) | 1st Intervention Period:Orlistat/Placebo (N=1) | 1st Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 1st Intervention Period:Orlistat/SLx-4090 (N=1) | 2nd Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=1) | 2nd Intervention Period:Orlistat/Placebo (N=1) | 2nd Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 2nd Intervention Period:Orlistat/SLx-4090 (N=2) | 3rd Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=1) | 3rd Intervention Period:Orlistat/Placebo (N=1) | 3rd Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 3rd Intervention Period:Orlistat/SLx-4090 (N=0) | 4th Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=1) | 4th Intervention Period:Orlistat/Placebo (N=0) | 4th Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 4th Intervention Period:Orlistat/SLx-4090 (N=0)
Pancreatitis. (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=2) | 1st Intervention Period:Orlistat/Placebo (N=1) | 1st Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 1st Intervention Period:Orlistat/SLx-4090 (N=1) | 2nd Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=1) | 2nd Intervention Period:Orlistat/Placebo (N=1) | 2nd Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 2nd Intervention Period:Orlistat/SLx-4090 (N=2) | 3rd Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=1) | 3rd Intervention Period:Orlistat/Placebo (N=1) | 3rd Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 3rd Intervention Period:Orlistat/SLx-4090 (N=0) | 4th Intervention Period:SLx-4090 Placebo/Orlistat Placebo (N=1) | 4th Intervention Period:Orlistat/Placebo (N=0) | 4th Intervention Period:Orlistat Placebo /Slx-4090 (N=1) | 4th Intervention Period:Orlistat/SLx-4090 (N=0)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased urgency of passing stool (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Only five patients were enrolled in the study. Two patients completed the study. One subject dropped our after Second Intervention Period. Participation of other two subjects was halted due to unavailability of study medications.

Study Design: Although protocol states "This trial is randomized, double-blind cross-over trial", study design was actually not a cross over design, but adaptive/flexible design using a responsive adaptive randomization. Thus Arm/Group were not listed "per sequence".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT01675154/Prot_SAP_000.pdf